CLINICAL TRIAL: NCT02779478
Title: Evaluation Of The Lung Microbiome In NTM Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01400
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Nontuberculous Mycobacteria; Bronchiectasis
Keywords: chronic obstructive pulmonary disease (COPD); cavitary; nodular bronchiectatic disease; NTM
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Airway microbiome using an aliquot of the induced sputum and upper airway samples. Since induced sputum may reflect different regions of the upper/lower airways, investigators will evaluate the upper and lower airway microbiome in a subgroup (case-control group) of patients using samples obtained through upper airway sampling and bronchoscopy, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive NTM Culture: Subjects that meet inclusion criteria and have culture positivity for NTM: at least two separate expectorated induced sputum samples or from one bronchoalveolar lavage (BAL) or lung biopsy
  Interventions: Procedure: Bronchoscopy
- Negative NTM Culture: Subjects that meet inclusion criteria and have less than two separate expectorated induced sputum samples culture negative or culture negative bronchoalveolar lavage (BAL) or lung biopsy.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy

SUMMARY:
A biomarker cohort study design is proposed to study whether specific airway microbiota alterations are associated with pulmonary Non-tuberculous mycobacteria (NTM) disease. In a cohort of 200 subjects suspected of having pulmonary NTM disease, the investigators will evaluate the airway microbiome using an aliquot of the induced sputum and upper airway samples. Since induced sputum may reflect different regions of the upper/lower airways, the investigators will evaluate the upper and lower airway microbiome in a subgroup (case-control group) of patients using samples obtained through upper airway sampling and bronchoscopy, respectively.

ELIGIBILITY:
Inclusion Criteria:

* History of pulmonary symptoms: cough, fatigue, malaise, fever, weight loss, dyspnea, hemoptysis, or chest discomfort
* Imaging abnormalities (within 2 years): defined as nodular or cavitary opacities on chest radiograph, or a computed tomography scan that shows bronchiectasis or bronchial wall thickening with associated multiple small nodules.

Definition of NTM case:

* Subjects that meet inclusion criteria and have culture positivity for NTM: at least two separate expectorated induced sputum samples or from one bronchoalveolar lavage (BAL) or lung biopsy

Definition of NTM control:

* Subjects that meet inclusion criteria and have less than two separate expectorated induced sputum samples culture negative or culture negative bronchoalveolar lavage (BAL) or lung biopsy.

Exclusion Criteria for cohort study (Aim 1-2):

* Recent (<1 months prior) oral antibiotic or steroid use. (Continuous treatment with macrolides and inhaled steroids are acceptable >1 month prior)
* Recent smoking history

Exclusion Criteria for bronchoscopic study (Aims 3-4):

* Forced expiratory volume at one second (FEV1) < 70%of predicted.
* Significant cardiovascular disease defined as abnormal EKG, known or suspected coronary artery disease or congestive heart failure.
* Diabetes mellitus
* Significant liver or renal disease
* Severe coagulopathy (INR > 1.4, Partial Thromboplastin Time (PTT) > 40 seconds and platelet count < 150x103 cells).
* Pregnancy
* Ethanol (ETOH) use of more than >6 beers or >4 mixed drinks daily
* Lack of capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Utilizing cohorts built at NYU over the last several years, this project is uniquely positioned to investigate the microbiome signatures among subjects with NTM disease.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of airway microbiome in subjects with active pulmonary NTM disease and compare with controls | 4 Hours
  Investigators will use sputum samples and brushed samples from areas of the upper airway from a cohort of 200 subjects with chronic cough and pulmonary infiltrates or airway abnormalities in whom NTM disease was suspected. Cultures positive for NTM (cases) will be compared to those with culture negatives (controls). Bacterial load by quantitative polymerase chain reaction (qPCR) will be used to characterize microbiome by high throughput sequencing looking for microbial biomarkers associated with NTM disease.

SECONDARY OUTCOMES:
Eating Assessment Tool (EAT-10) to evaluate the prevalence of laryngopharyngeal reflux and dysphagia/aspiration in subjects with active pulmonary NTM disease compared with controls | 1 Hour
Laryngoscopy to calculate the Reflux finding score (RFS, a validated quantitative measurement of impact of laryngopharyngeal reflux on the upper airway in adults | 4 Hours
Reflux Symptom Index evaluate the prevalence of laryngopharyngeal reflux and dysphagia/aspiration in subjects with active pulmonary NTM disease compared with controls | 1 Hour

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Segal, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States